CLINICAL TRIAL: NCT05518409
Title: Immunohistochemical Study of Peripheral Blood Mononuclear Cells in Sporadic Alzheimer's Disease and Dementia With Lewy Body
Brief Title: Immunohistochemical Study of Neurodegenerative Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Hu ShaoHua, Department of Psychiatry, First Affiliated Hospital of Zhejiang University, First Affiliated Hospital of Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IIT20220213B-R1
Record Dates: First submitted 2022-08-09; First posted 2022-08-26 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Alzheimer Disease; Lewy Body Disease; Neurodegenerative Diseases
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Neurodegenerative Diseases | interventions — Donepezil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AD group (Experimental): 20 subjects who met the diagnostic criteria and exclusion criteria of AD were included in the discovery cohort.
  Interventions: Biological: Detection of cytof in peripheral PBMC; Drug: Donepezil for patients with AD and DLB
- DLB group (Experimental): Of the 30 subjects who met the DLB diagnostic criteria and exclusion criteria, 20 were included in the discovery cohort and 10 in the validation cohort.
  Interventions: Biological: Detection of cytof in peripheral PBMC; Drug: Donepezil for patients with AD and DLB
- Healthy control group (Experimental): Among the 30 subjects who met the diagnostic and exclusion criteria of the healthy control group, 20 were included in the discovery cohort and 10 in the validation cohort.
  Interventions: Biological: Detection of cytof in peripheral PBMC

INTERVENTIONS:
Biological: Detection of cytof in peripheral PBMC — Each subject needs to take 5ml of peripheral venous blood to extract PBMC cells, and then conduct cytof detection. This is a mass spectrometry flow cytometry method based on single cell level. It has the ability to analyze all immune cells with high resolution.
Drug: Donepezil for patients with AD and DLB — The subjects in AD and DLB groups were given donepezil at an initial dose of 5mg and then increased to 10mg one month later. Lasting for 1 year.
  Arms: AD group; DLB group

SUMMARY:
The subject uses cytof to analyze PBMC of sporadic AD and DLB, which is used to reveal the differences in immune characteristics of the two diseases at the single-cell level, build immune models for specific diseases, and define these two neurodegenerative diseases with high precision from the level of molecular immunity. To provide basis for further study of the immunohistochemical differences between the two diseases, and provide objective support for clinical diagnosis and differential diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. AD inclusion criteria:

   a.Clinical diagnosis of Alzheimer's Disease
2. DLB inclusion criteria:

   1. Clinical diagnosis of Dementia with Lewy bodies

Exclusion Criteria:

1. Infectious diseases
2. autoimmune disease
3. heart failure
4. chronic obstructive pulmonary disease (COPD)
5. cancer
6. renal failure
7. recently major surgery
8. alcohol and / or drug abuse
9. disturbance of consciousness
10. clinical diagnosis of major depression disorder
11. clinical diagnosis of Anxiety disorder

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Immunerepertorie | 1 year
  The immune cells were drawn into immunoreceptor by mass cytometry (cytof) technology. Immunerepertorie is used for the classification of immune cells. According to the proportion of various immune cell subtypes and biomarkers in all cells, it is used to find the difference between immune cell subtypes and biomarkers in different diseases. Scoring frame: 0-1. The higher the score, the greater the proportion of this subtype or biomarker.
immunological Elastic-Net (iEN) model | 1 year
  The immunological Elastic-Net (iEN), which incorporates immunological knowledge directly into the predictive models. The ROC curve output by the model is plotted with specificity as the abscissa and sensitivity as the ordinate, and the AUC (area under the curve) value is calculated. The AUC value was used to evaluate the authenticity of the IEN model. Score frame: 0.5-1. A higher value indicates that the model is closer to the real situation.

SECONDARY OUTCOMES:
Mini-mental State Examination（MMSE） | 1 year
  MMSE was used to evaluate the degree of intellectual status and cognitive impairment. Score frame: 0 ~ 30. The lower the score, the more severe the cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Li YouMing, Study Chair — Zhejiang University
Locations (1):
- Department of Psychiatry, First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China